CLINICAL TRIAL: NCT01609738
Title: Left Ventricular Septum Pacing in Patients by Transvenous Approach Through the Inter-ventricular Septum - Feasibility, Long-term Lead Stability and Safety
Brief Title: Left Ventricular Septum Pacing in Patients by Transvenous Approach Through the Inter-ventricular Septum
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: NL37648.068.11; METC 11-1-047 (Other: METC azm/UM)
Record Dates: First submitted 2012-04-05; First posted 2012-06-01 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Left Ventricular Dysfunction; Cardiac Conduction Defect; Heart Failure; Sick Sinus Syndrome
Keywords: Cardiac pacing; Left ventricular septal pacing; Feasibility and safety; Lead stability; Hemodynamics; Left ventricular dyssynchrony; Pacing for heart failure; Cardiac resynchronization therapy
MeSH Terms: conditions — Ventricular Dysfunction, Left; Cardiac Conduction System Disease; Heart Failure; Sick Sinus Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sinus node dysfunction: Patients with sinus node dysfunction and structurally normal hearts
  Interventions: Device: Left ventricular septum pacing lead
- CRT indication: Patients with an indication for CRT (heart failure with an LVEF <35% and LBBB)
  Interventions: Device: Left ventricular septum pacing lead

INTERVENTIONS:
Device: Left ventricular septum pacing lead — A left ventricular septum pacing lead is permanently placed by introducing a custom lead with extended helix transvenously and, after positioning it against the RV septum, driving it through the inter-ventricular septum into the LV endocardial layer.
  Other Names: Adapted Medtronic Select Secure 3830 pacing lead

SUMMARY:
Cardiac pacing is the only effective treatment for symptomatic bradycardia. The right ventricular apex (RVA) has become the most frequently used ventricular pacing site. However, RVA pacing has been shown to cause left ventricular (LV) dyssynchrony wich can lead to LV dysfunction and development of heart failure. Recent studies in animals have demonstrated that pacing at the LV septum induces significantly less ventricular dyssynchrony than RVA pacing and is able to improve LV function to a similar degree as biventricular (BiV) pacing. In addition it was shown that a LV septum lead can be placed permanently by driving a lead with extended helix from the RV side through the inter-ventricular septum into the LV endocardial layer. This was shown to be a feasible and safe procedure and lead stability was shown during four months of follow-up in otherwise healthy and active canines. LV septum pacing may therefore be a good treatment alternative in patients with symptomatic bradycardia, as well as patients with an indication for cardiac resynchronization therapy (CRT). The purpose of this study is to translate the findings from preclinical studies to the clinical situation by investigating the feasibility, long-term lead stability and safety of LV septum pacing by transvenous approach through the inter-ventricular septum in patients.

DETAILED DESCRIPTION:
Cardiac pacing is the only effective treatment for symptomatic bradycardia. After the introduction of the implantable pacemaker (PM), the right ventricular apex (RVA) has become the most frequently used ventricular pacing site. However, clinical studies have shown that RVA pacing leads to left ventricular (LV) dyssynchrony, and on the long run to adverse structural changes (remodeling), a higher risk of developing atrial fibrillation and heart failure, and higher mortality.

Recognition of the adverse effects of RVA pacing has generated interest in alternative ventricular pacing sites. Recent studies in animals have shown that pacing at the LV septum induces significantly less ventricular dyssynchrony than RVA pacing. In addition it was shown that a LV septum lead can be placed permanently by introducing a custom lead with extended helix transvenously and, after positioning it against the RV septum, driving it through the inter-ventricular septum into the LV endocardial layer. This was shown to be a feasible and safe procedure and lead stability was shown during four months of follow-up in otherwise healthy and active canines.

Animal studies have also shown that LV septum pacing is able to improve LV function to a similar degree as simultaneous biventricular (BiV) pacing used in cardiac resynchronization therapy (CRT). CRT was introduced to restore the abnormal ventricular activation and contraction in patients with heart failure and intra-ventricular conduction delay. Large clinical trials have shown that CRT improves LV systolic pump function, reverses structural remodelling, improves quality of life and exercise tolerance, and decreases mortality. Unfortunately, problems encountered during positioning and fixation of the LV pacing lead in the coronary vein result in suboptimal or loss of CRT in at least a quarter of CRT candidates and require re-operation in 7% during follow up.

The adverse effects of RVA pacing, the limitations of BiV pacing and the promising effects of LV septum pacing in preclinical studies have led to the idea that LV septum pacing may be a good treatment alternative in patients with symptomatic bradycardia, as well as patients with an indication for CRT. In the latter category, CRT could then be performed using a single ventricular pacing lead, thus limiting the number of lead implantations, and thereby reducing complication rate and implantation costs as well as avoiding the difficult access route through the coronary vein.

It is the aim of this study to translate the findings from preclinical studies to the clinical situation by investigating the feasibility, long-term lead stability and safety of LV septum pacing by transvenous approach through the inter-ventricular septum in patients with a PM or CRT indication. The results may have a large impact on future pacing therapy. The LV septum may become the universal pacing site, being preferred for anti-bradycardia therapy, and being an equal alternative for BiV pacing, but easier to apply, less invasive and more cost-effective.

ELIGIBILITY:
Inclusion Criteria:

1. Cardiac pacing indication for sinus node dysfunction (dual chamber pacemaker) or indication for CRT (BiV pacemaker).

   * Patient with sinus node dysfunction:
   * Normal left ventricular ejection fraction (LVEF > 50%)
   * Left ventricular end-diastolic diameter (LVEDD) < 55mm
   * QRS duration < 100ms
   * Patient with CRT indication:
   * Non-ischemic cardiomyopathy
   * LVEF is < 35%
   * Typical left bundle-branch block on surface ECG
   * QRS duration >150ms
   * NYHA functional class I-III
2. Greater than 18 years of age
3. Stable sinus rhythm at the time of inclusion
4. Willing and capable of giving informed consent

Exclusion Criteria:

1. Ventricular pacing dependent
2. High degree AV block
3. Previous septal myocardial infarction
4. Previously implanted pacing device
5. Abnormal venous anatomy
6. Left ventricular septum wall thickness >10mm determined by echocardiography
7. Presence of severe valvular disease
8. Presence of an ongoing progressive terminal disease associated with a reduced likelihood of survival for the duration of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects are recruited from patients referred to the out-patient pacemaker/ICD clinic of our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of successful LV septum lead implantations | Baseline and 6 months
  LV septum lead implantation is considered successful if the lead can be placed in the endocardial LV septum and adequate and stable sensing and pacing tresholds are achieved.
Change in sensing values, pacing threshold and lead impedance | Baseline and 6 months
  Maintenance of stable lead function is determined by assessment of change in the electrical parameters: sensing value, pacing threshold and lead impedance at baseline versus 6 months follow-up.
Number of participants with procedure or lead related adverse events | Baseline and 6 months
  The number of participant with and the kind of procedure- or lead related complications are assessed at the time of the procedure and up to 6 months after lead implantation. Special attention is given to the presence of perforation or rupture of the inter-ventricular septum or free wall, pericardial effusion, thrombosis, heart rhythm disturbances, conduction disturbances, and lead-/screw dislocation/-fracture.

SECONDARY OUTCOMES:
Acute change in LVdP/dtmax | Acute measurements are performed for the duration of the lead implantation procedure, an expected average of two hours
  Acute change in LV systolic function using the hemodynamic parameter LVdP/dtmax during LV septum pacing compared to:
  * RVA pacing and baseline (atrial pacing / AAI mode) in patients with SND.
  * RVA pacing, single LV epicardial lateral wall pacing, Bi-LV pacing (LV septum and LV lateral wall pacing), BiV pacing (RV septum and LV lateral wall pacing) and baseline (atrial pacing / AAI mode) in heart failure patients who are candidates for CRT.
Acute change in LV stroke volume | Acute measurements are performed for the duration of the lead implantation procedure, an expected average of two hours
  Acute change in LV systolic function using the hemodynamic parameter LV stroke volume measured by Nexfin, during LV septum pacing compared to:
  * RVA pacing and baseline (atrial pacing / AAI mode) in patients with SND.
  * RVA pacing, single LV epicardial lateral wall pacing, Bi-LV pacing (LV septum and LV lateral wall pacing), BiV pacing (RV septum and LV lateral wall pacing) and baseline (atrial pacing / AAI mode) in heart failure patients who are candidates for CRT.
Acute change in QRS duration | Baseline and 4 weeks
  Acute change in sequence of LV electrical activation using the electrocardiographic parameter QRS duration, during LV septum pacing compared to:
  * RVA pacing and baseline (atrial pacing / AAI mode) in patients with SND.
  * RVA pacing, single LV epicardial lateral wall pacing, Bi-LV pacing (LV septum and LV lateral wall pacing), BiV pacing (RV septum and LV lateral wall pacing) and baseline (atrial pacing / AAI mode) in heart failure patients who are candidates for CRT.
Acute change in 3-dimensional QRS vector direction | Baseline and 4 weeks
  Acute change in sequence of LV electrical activation using the electrocardiographic parameter 3-dimensional QRS vector direction, during LV septum pacing compared to:
  * RVA pacing and baseline (atrial pacing / AAI mode) in patients with SND.
  * RVA pacing, single LV epicardial lateral wall pacing, Bi-LV pacing (LV septum and LV lateral wall pacing), BiV pacing (RV septum and LV lateral wall pacing) and baseline (atrial pacing / AAI mode) in heart failure patients who are candidates for CRT.
Acute change in SPECKLE-tracking strain | Baseline and 4 weeks
  Acute change in regional myocardial deformation patterns using the echocardiographic parameter SPECKLE-tracking strain, during LV septum pacing compared to:
  * RVA pacing and baseline (atrial pacing / AAI mode) in patients with SND.
  * RVA pacing, single LV epicardial lateral wall pacing, Bi-LV pacing (LV septum and LV lateral wall pacing), BiV pacing (RV septum and LV lateral wall pacing) and baseline (atrial pacing / AAI mode) in heart failure patients who are candidates for CRT.
Difference between relative changes in LV stroke volume assessed by Nexfin and relative changes in invasively measured LVdp/dtmax. | Acute measurements are performed for the duration of the lead implantation procedure, an expected average of two hours
  Correlation between the relative change in non-invasively measured LV stroke volume using Nexfin and the relatieve change in invasively determined LV dP/dtmax, during LV septum pacing compared to:
  * RVA pacing and baseline (atrial pacing / AAI mode) in patients with SND.
  * RVA pacing, single LV epicardial lateral wall pacing, Bi-LV pacing (LV septum and LV lateral wall pacing), BiV pacing (RV septum and LV lateral wall pacing) and baseline (atrial pacing / AAI mode) in heart failure patients who are candidates for CRT.

CONTACTS AND LOCATIONS:
Overall Officials: Frits Prinzen, PhD, Principal Investigator — Maastricht University; Kevin Vernooy, MD, PhD, Study Director — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Mills RW, Cornelussen RN, Mulligan LJ, Strik M, Rademakers LM, Skadsberg ND, van Hunnik A, Kuiper M, Lampert A, Delhaas T, Prinzen FW. Left ventricular septal and left ventricular apical pacing chronically maintain cardiac contractile coordination, pump function and efficiency. Circ Arrhythm Electrophysiol. 2009 Oct;2(5):571-9. doi: 10.1161/CIRCEP.109.882910. Epub 2009 Aug 25. PMID 19843926
- [Background] Peschar M, de Swart H, Michels KJ, Reneman RS, Prinzen FW. Left ventricular septal and apex pacing for optimal pump function in canine hearts. J Am Coll Cardiol. 2003 Apr 2;41(7):1218-26. doi: 10.1016/s0735-1097(03)00091-3. PMID 12679225
- [Background] Grosfeld MJ, Res JC, Vos DH, de Boer TJ, Bos HJ. Testing a new mechanism for left interventricular septal pacing: the transseptal route; a feasibility and safety study. Europace. 2002 Oct;4(4):439-44. doi: 10.1053/eupc.2002.0253. PMID 12408265
- [Background] Andersen HR, Nielsen JC, Thomsen PE, Thuesen L, Mortensen PT, Vesterlund T, Pedersen AK. Long-term follow-up of patients from a randomised trial of atrial versus ventricular pacing for sick-sinus syndrome. Lancet. 1997 Oct 25;350(9086):1210-6. doi: 10.1016/S0140-6736(97)03425-9. PMID 9652562
- [Background] Wilkoff BL, Cook JR, Epstein AE, Greene HL, Hallstrom AP, Hsia H, Kutalek SP, Sharma A; Dual Chamber and VVI Implantable Defibrillator Trial Investigators. Dual-chamber pacing or ventricular backup pacing in patients with an implantable defibrillator: the Dual Chamber and VVI Implantable Defibrillator (DAVID) Trial. JAMA. 2002 Dec 25;288(24):3115-23. doi: 10.1001/jama.288.24.3115. PMID 12495391
- [Background] Sweeney MO, Hellkamp AS, Ellenbogen KA, Greenspon AJ, Freedman RA, Lee KL, Lamas GA; MOde Selection Trial Investigators. Adverse effect of ventricular pacing on heart failure and atrial fibrillation among patients with normal baseline QRS duration in a clinical trial of pacemaker therapy for sinus node dysfunction. Circulation. 2003 Jun 17;107(23):2932-7. doi: 10.1161/01.CIR.0000072769.17295.B1. Epub 2003 Jun 2. PMID 12782566
- [Background] Lamas GA, Lee KL, Sweeney MO, Silverman R, Leon A, Yee R, Marinchak RA, Flaker G, Schron E, Orav EJ, Hellkamp AS, Greer S, McAnulty J, Ellenbogen K, Ehlert F, Freedman RA, Estes NA 3rd, Greenspon A, Goldman L; Mode Selection Trial in Sinus-Node Dysfunction. Ventricular pacing or dual-chamber pacing for sinus-node dysfunction. N Engl J Med. 2002 Jun 13;346(24):1854-62. doi: 10.1056/NEJMoa013040. PMID 12063369
- [Background] Steinberg JS, Fischer A, Wang P, Schuger C, Daubert J, McNitt S, Andrews M, Brown M, Hall WJ, Zareba W, Moss AJ; MADIT II Investigators. The clinical implications of cumulative right ventricular pacing in the multicenter automatic defibrillator trial II. J Cardiovasc Electrophysiol. 2005 Apr;16(4):359-65. doi: 10.1046/j.1540-8167.2005.50038.x. PMID 15828875
- [Background] Auricchio A, Stellbrink C, Block M, Sack S, Vogt J, Bakker P, Klein H, Kramer A, Ding J, Salo R, Tockman B, Pochet T, Spinelli J. Effect of pacing chamber and atrioventricular delay on acute systolic function of paced patients with congestive heart failure. The Pacing Therapies for Congestive Heart Failure Study Group. The Guidant Congestive Heart Failure Research Group. Circulation. 1999 Jun 15;99(23):2993-3001. doi: 10.1161/01.cir.99.23.2993. PMID 10368116
- [Background] Wecke L, Rubulis A, Lundahl G, Rosen MR, Bergfeldt L. Right ventricular pacing-induced electrophysiological remodeling in the human heart and its relationship to cardiac memory. Heart Rhythm. 2007 Dec;4(12):1477-86. doi: 10.1016/j.hrthm.2007.08.001. Epub 2007 Aug 11. PMID 17997360